CLINICAL TRIAL: NCT03070964
Title: A Phase II Study of Plitidepsin in Patients With Relapsed or Refractory Angioimmunoblastic T-cell Lymphoma
Brief Title: A Study of Plitidepsin in Patients With Relapsed or Refractory Angioimmunoblastic T-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The main reason that motivated the study termination was the slow recruitment of the trial.
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-B-021-13
Record Dates: First submitted 2017-01-16; First posted 2017-03-06 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — plitidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plitidepsin (Experimental)
  Interventions: Drug: plitidepsin

INTERVENTIONS:
Drug: plitidepsin
  Other Names: APLD Aplidine

SUMMARY:
Prospective, multicenter, phase II clinical trial to determine the efficacy of plitidepsin in patients with relapsed/refractory (R/R) angioimmunoblastic Tcell lymphoma (AITL).This is an international, multicenter study (with approximately 17 investigative sites).

DETAILED DESCRIPTION:
Prospective, multicenter, phase II clinical trial to determine the efficacy of plitidepsin in patients with relapsed/refractory (R/R) AITL. The primary endpoint will be overall response rate (ORR) according to the Lugano classification response criteria per independent review.

Medical specialists (radiologists and hematologists) who are directly involved in the care of patients with AITL (but are not participating in this trial as investigators) will review all efficacy data (including radiological assessments, bone marrow biopsies) and will assign the best response and the date of objective response or progression/censoring according to their independent evaluation.

Central pathological review of each patient's original diagnosis report(s) will be required before inclusion.

Two futility analyses of the primary endpoint (ORR according to the Lugano classification criteria and per Independent Review Committee (IRC)) are planned around six months after approximately 25% and 50% of eligible patients (i.e., 15 and 30 patients respectively with AITL confirmed by central pathological review) have been treated. Two or less responders out of 15 patients or seven or less responders out of 30 patients, according to boundaries and sample size assumptions, will mean that the alternative hypothesis could be rejected, and thus recruitment might be stopped at the time of the first or second futility analysis, respectively. Otherwise, accrual will continue to 60 patients with AITL confirmed by central pathological review. This decision will be taken at the time by an Independent Data Monitoring Committee (IDMC). The IDMC, which will include specialists in peripheral T-cell lymphomas (PTCL) supported by a medical statistician, will review data provided by the Investigators, the IRC efficacy assessments and safety information and will advise whether the study should continue. Recruitment can continue during the review period.

If there are 19 or more responders of 60 patients, the efficacy of plitidepsin will be considered as clinically relevant in AITL patients.

Central pathological review will be conducted by experienced pathologists appointed by the Sponsor and available to the investigative sites for consultation about AITL diagnosis confirmation. Central pathological review is required for (a) local histopathology reports prior to patient treatment, and (b) tumor samples before each futility analysis and at the end of the study.

The central laboratory pathologists will be responsible for (a) approving patient inclusion on the basis of investigative site pathology reports provided during screening, (b) analyzing tumor biopsies (initial diagnosis and/or relapses) to confirm the AITL diagnosis, and (c) analyzing blood samples to identify plasma biomarkers and extract DNA.

Tumor samples (initial diagnosis and relapses) are required for central review to confirm AITL diagnosis but not to approve inclusion. Archived tissue samples of representative tumors must be sent for central review and biomarker analysis. If the diagnosis biopsy is not available (because the patient was diagnosed at another site, for example), the most recent representative biopsy (relapse and/or progression) will be used. Submitting both, however, is strongly recommended. Tumor blocks will be returned to the centers.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the patient (both to participate in the study and to provide biopsy samples) obtained before any study-specific procedure.
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
4. Life expectancy ≥ 3 months.
5. Histologically confirmed diagnosis of R/R AITL (eligibility needs to be confirmed by central pathological review).
6. At least a two-week washout period since the end of the last therapy (six weeks for a prior nitrosourea-containing regimen), recovery to grade ≤ 1 from any non-hematological adverse event (AE) derived from previous treatment (excluding alopecia).
7. Adequate bone marrow (BM), renal, hepatic, and metabolic function (assessed ≤ 14 days before inclusion in the study):

   1. Absolute neutrophil count (ANC) ≥ 1.0 × 109/L. Screening of ANC should be independent of granulocytecolony stimulating factor (G-CSF) support for at least one week and of pegylated G-CSF for at least two weeks.
   2. Platelet count ≥ 75 × 109/L.
   3. Hemoglobin ≥ 9 g/dL. Patients may receive red blood cells (RBC) and/or erythropoietin (EPO) and/or platelet transfusions in accordance with institutional guidelines.
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × the upper limit of normal (ULN).
   5. Total bilirubin ≤ 1.5 × ULN.
   6. Alkaline phosphatase (ALP) ≤ 3.0 × ULN (< 5 × ULN if isolated ALP increase, i.e., without ALT/AST or bilirubin increase).
   7. Calculated creatinine clearance (CrCL) ≥ 30 mL/minute (Cockcroft-Gault formula).
   8. Creatine phosphokinase (CPK) ≤ 2.5 × ULN.
   9. Albumin ≥ 2.5 g/dL.
8. Left ventricular ejection fraction (LVEF) by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan within normal range (according to institutional standards).

Exclusion Criteria:

1. Prior treatment with plitidepsin.
2. Concomitant diseases/conditions:

   1. History or presence of angina, myocardial infarction, clinically relevant valvular heart disease, uncontrolled hypertension, or congestive heart failure within the previous 12 months.
   2. Symptomatic arrhythmia (excluding grade ≤ 2 anemia-related sinusal tachycardia) or any arrhythmia requiring ongoing treatment, and/or prolonged grade ≥ 2 QT-QTc, or presence of unstable atrial fibrillation. Patients with stable atrial fibrillation on treatment are allowed provided they do not meet any other cardiac or prohibited drug exclusion criterion.
   3. Active uncontrolled infection. Active hepatitis B or C virus (HBV or HCV), or human immunodeficiency virus (HIV)infection.
   4. Morphological or cytological features of myelodysplasia and/or post chemotherapy aplasia on bone marrow (BM) assessment.
   5. Myopathy > grade 2 or any clinical situation that causes significant and persistent elevation of CPK (> 2.5 × ULN in two different determinations performed one week apart).
   6. Limitation of the patient's ability to comply with the treatment or follow-up requirements.
   7. Diagnosis of another invasive malignancy unless free of disease for at least three years following therapy with curative intent. Patients with early-stage basal cell or squamous cell skin cancer, cervical intraepithelial neoplasia, cervical carcinoma in situ, or superficial bladder cancer, may be eligible to participate at the Investigator's discretion.
   8. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
3. Central nervous system (CNS) involvement.
4. Women who are pregnant or breast feeding. Fertile patients (men and women) who are not using an effective method of contraception. All patients (men and women) must agree to use an effective contraceptive measure (if applicable) up to six months after treatment discontinuation.
5. Concomitant medications that include corticosteroids, chemotherapy, or other therapy that is or may be active against AITL, within the two weeks prior to treatment start. Concurrent corticosteroids are allowed, provided they are administered at an equivalent prednisone dose of ≤ 10 mg daily, as premedication for blood products only.
6. Major upper gastrointestinal bleeding episode occurring during the previous year before screening.
7. Known hypersensitivity to any of plitidepsin's formulation components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (2):
  - Northwestern University Medical School, Chicago, Illinois
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Czechia (2):
  - Faculty Hospital Ostrava, Ostrava
  - Fakultni Nemocnice Praha, Prague
- Italy (4):
  - Ospedale Clinico Aviano, Aviano, Pordenone
  - Instituto di Ematologia "Seragnoli", Bologna
  - Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria Careggi, Florence
- Spain (9):
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Centro Oncológico MD Anderson International España, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen del Rocío, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first IC was signed on 25Oct2016 and the first study treatment administration was on 9Nov2016.
  The cutoff date was 2Jul2018 (date of last follow-up, clinical cutoff). At cutoff date, 14 patients had been included, of whom 13 were treated and evaluable for safety, and 12 were evaluable for the primary efficacy endpoint
Groups:
- Plitidepsin: Plitidepsin was administered i.v. as a 1-hour infusion (fixed rate) via central or peripheral venous catheter. Patients received plitidepsin at a starting dose of 3.2 mg/m2 on Day 1, 8 and 15 every four weeks (q4wk). A 1-day window is allowed for plitidepsin administration. A cycle is defined as a fourweek period. A 1-day window was allowed for plitidepsin administration.
Period: Overall Study
Arm/Group | Plitidepsin
Started | 14
Completed | 0
Not Completed | 14
Not completed — Progressive disease | 8
Not completed — Treatment-unrelated adverse event | 2
Not completed — Never treated | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Plitidepsin
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 61 [40 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13
  Hispanolatin | 1
ECOG PS [Count of Participants; unit: Participants] — ECOG PS, Eastern Cooperative Oncology Group performance status PS 0 Fully active able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities up and about more than 50% of waking hours PS 3 Capable of only limited selfcare confined to bed or chair more than 50% of waking hours PS 4 Completely disabled cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    PS 0 | 8
    PS 1 | 5
    PS 2 | 1
Ann Arbor stage [Count of Participants; unit: Participants] — Stages:
  I cancer in a single region, usually one lymph node and the surrounding area. No outward symptoms II cancer in 2 separate regions, an affected lymph node or lymphatic organ and a 2nd affected area. Both affected areas are confined to one side of the diaphragm III cancer has spread to both sides of the diaphragm, including one organ or area near the lymph nodes or the spleen IV disseminated involvement of one/more extralymphatic organs A/B the absence of constitutional B-type symptoms is denoted by adding an A to stage; the presence adding a B
  Participants
    III | 1
    III-A | 3
    III-B | 3
    IV-A | 3
    IV-B | 4
Extranodal disease at diagnosis [Count of Participants; unit: Participants]
  Yes | 5
  No | 9
Bulky lesion at diagnosis [Count of Participants; unit: Participants]
  Yes | 1
  No | 13
International Prognostic Index score at diagnosis [Count of Participants; unit: Participants]
  Low risk (0-1 risk factors) | 2
  Low-intermediate risk (2 risk factors) | 2
  High-intermediate risk (3 risk factors) | 2
  High risk (4-5 risk factors) | 4
  NA | 4
Prognostic index for peripheral T-cell lymphoma at diagnosis [Count of Participants; unit: Participants]
  Group 1 (no adverse factors) | 1
  Group 2 (1 risk factor) | 1
  Group 4 (3-4 risk factors) | 2
  NA | 10
Prognostic index for angioimmunoblastic T-cell lymphoma score at diagnosis [Count of Participants; unit: Participants]
  Low-risk group | 3
  High-risk group | 3
  NA | 8
International prognostic index score at current disease [Count of Participants; unit: Participants]
  Low risk (0-1 risk factors) | 3
  Low-intermediate risk (2 risk factors) | 3
  High-intermediate risk (3 risk factors) | 4
  High risk (4-5 risk factors) | 4
Prognostic index for peripheral T-cell lymphoma at current disease [Count of Participants; unit: Participants]
  Group 1 (no adverse factors) | 2
  Group 2 (1 risk factor) | 3
  Group 3 (2 risk factors) | 1
  Group 4 (3-4 risk factors) | 1
  NA | 7
Prognostic index for angioimmunoblastic T-cell lymphoma score at current disease [Count of Participants; unit: Participants]
  Low-risk group | 5
  High-risk group | 4
  NA | 5
Prior anticancer therapy lines [Count of Participants; unit: Participants]
  1 line | 2
  2 lines | 5
  3 lines | 5
  4 lines | 1
  5 lines | 1
Best response to last prior therapy [Count of Participants; unit: Participants] — CR, complete response; PD, disease progression; PR, partial response; SD, stable disease; UK, unknown
  Participants
    CR | 4
    PR | 4
    SD | 1
    PD | 3
    UK | 2
Prior stem cell transplantation [Count of Participants; unit: Participants]
  NO | 8
  Allogenic stem cell transplantation | 1
  Autologous stem cell transplantation | 5
Weight [Median (Full Range); unit: Kg] | 72.5 [44.7 to 145.0]
Height [Median (Full Range); unit: cm] | 166.5 [152 to 190]
Body Surface Area [Median (Full Range); unit: m^2] | 1.8 [1.4 to 2.8]
Time from diagnosis to first plitidepsin infusion [Median (Full Range); unit: months] | 24.1 [8.5 to 200.5]
Time from last progressive disease to infusion [Median (Full Range); unit: weeks] | 6.9 [0.9 to 54.0]
Prior anticancer therapy lines [Median (Full Range); unit: therapy lines] | 2.5 [1 to 5]
Time to progressions to last anticancer therapy [Median (Full Range); unit: months] | 4.6 [1.5 to 92.5]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate by the Lugano Classification Per Independent Review Assessment
Description: The study protocol established that the analysis of the primary endpoint should have been done once a total of 60 patients have received plitidepsin, with two futility analyses planned after the inclusion of approximately 15 and 30 patients, respectively. However, only a total of 14 patients were included, of whom 13 were treated, and 12 were evaluable for the primary efficacy endpoint (ORR per IRC in the "Per Protocol Patients" population). As a result of slow patient accrual, the study was closed before reaching the target enrollment of 15 patients for the first futility analysis, and the primary endpoint (ORR according to the Lugano classification criteria and per IRC) was not assessed.
Time Frame: Change from Baseline to assessments at: 1/2 weeks after cycle 3 and 4-8 weeks after cycle 6 (1cycle =28days), follow-up every 4 months +/- 2 weeks until progression disease or end of study (expected: 42 months)
Population: Justification: The study was closed before reaching the target enrollment of 15 patients for the first futility analysis, and the primary endpoint (ORR according to the Lugano classification criteria and per IRC) was not assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Plitidepsin
Number analyzed (Participants) | 12
Participants | NA — ORR according to the Lugano classification criteria per IRC was not assessed

2. Secondary Outcome: Overall Response Rate by Investigator's Assessment - Per Protocol Patients Population
Description: CI, confidence interval; CR, complete response; NE, not evaluable; ORR, overall response rate; PD, disease progression; PR, partial response; SD, stable disease.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From the date when the remission criteria are fulfilled to the first date when progressive disease, recurrence or death (due to any cause)is documented, expected at a maximum of 42 months
Population: A patient was never treated with plitidepsin. A patient due to lack of AITL diagnosis confirmation
Measure: Count of Participants; unit: Participants
Arm/Group | Plitidepsin
Number analyzed (Participants) | 12
Participants
  CR | 1
  PR | 1
  SD | 1
  PD | 7
  NE | 2
Statistical Analysis 1: Comparison: Plitidepsin; Test type: Superiority; Exact binomial estimator = 16.7, 95% CI 2-sided [2.1 to 48.4]

ADVERSE EVENTS:
Time Frame: Participants were assessed through study completion, approximately 2 years
Description: One patient was never treated with plitidepsin and was excluded from the analysis of safety.
Arm/Group | Plitidepsin
All-Cause Mortality (participants affected / at risk) | 7/13
Serious Adverse Events (participants affected / at risk) | 9/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plitidepsin (N=13)
Peripheral embolism (Vascular disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Rhinovirus infection (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plitidepsin (N=13)
Subclavian vein thrombosis (Vascular disorders) | 1 (1)
Asthenia/Fatigue (General disorders) | 4 (6)
Chills (General disorders) | 1 (2)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 3 (3)
Pyrexia (General disorders) | 6 (17)
Insomnia (Psychiatric disorders) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (15)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (6)
Weight decreased (Investigations) | 1 (1)
Anaemia (Investigations) | 3 (13)
Eosinophilia (Investigations) | 1 (1)
Lymphadenopathy (Investigations) | 1 (1)
Neutropenia (Investigations) | 2 (2)
Thrombocytopenia (Investigations) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysaesthesia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (7)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastric mucosa erythema (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 3 (8)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2)
Rhinovirus infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
On 14May18, Sponsor informed to the sites and IPs its decision to close the recruitment. Study was terminated before reaching the target enrollment due to slow patient accrual and the negative opinion of the EMA-refusal of the mark. auth. plitidepsin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT03070964/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03070964/SAP_001.pdf